CLINICAL TRIAL: NCT07172269
Title: Evaluation the Effect of Mangosteen Supplement as Adjuvant Therapy With Sitagliptin/Metformin in Type 2 Diabetic Iraqi Patients
Brief Title: Mangosteen Supplement as Adjuvant Therapy With Sitagliptin/Metformin in Iraqi Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mais Qais Hbeeb (Other)
Responsible Party: Sponsor-Investigator, Mais Qais Hbeeb, MSC Candidate, department of clinical pharmacy , college of pharmacy, Mustansiriyah university, Baghdad, Iraq, Al-Mustansiriyah University
Organization: Al-Mustansiriyah University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 92
Record Dates: First submitted 2025-09-06; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Diabete Mellitus; Type 2 Diabetes; Obesity Type 2 Diabetes Mellitus; Dyslipidemia in Patients With Diabetes Mellitus; Insulin Resistance
Keywords: Diabetes Mellitus; Diabete Type 2; T2DM; Mangosteen; sitagliptin; metformin; xanthones; antioxidant; inflammation
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Insulin Resistance; Inflammation | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Intervention Model Description: Participants were randomized into two parallel groups. Group 1 received sitagliptin/metformin (50/1000 mg twice daily) plus lifestyle modification. Group 2 received sitagliptin/metformin (50/1000 mg twice daily) plus mangosteen supplement (500 mg twice daily) with lifestyle modification. The intervention period lasted 12 weeks.
Masking Description: This is open-label study, no parties were masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitagliptin/Metformin + Lifestyle Modification (Active Comparator): Patients receive sitagliptin/metformin tablets (50/1000 mg) orally, twice daily for 12 weeks, in addition to lifestyle modification including diet counseling, exercise, and diabetes education.
  Interventions: Drug: Sitagliptin + Metformin; Behavioral: Lifestyle Management
- Sitagliptin/Metformin + Mangosteen + Lifestyle Modification (Experimental): Patients receive sitagliptin/metformin tablets (50/1000 mg) orally, twice daily, plus mangosteen capsules (500 mg) orally, twice daily for 12 weeks, in addition to lifestyle modification including diet counseling, exercise, and diabetes education.
  Interventions: Drug: Sitagliptin + Metformin; Dietary Supplement: mangosteen supplement; Behavioral: Lifestyle Management

INTERVENTIONS:
Drug: Sitagliptin + Metformin — Oral tablets, 50/1000 mg, taken twice daily after meals for 12 weeks
  Other Names: Sitadin M
Dietary Supplement: mangosteen supplement — Capsules, 500 mg, taken twice daily after meals for 12 weeks
  Other Names: Garcinia mangostana extract
  Arms: Sitagliptin/Metformin + Mangosteen + Lifestyle Modification
Behavioral: Lifestyle Management — Diabetes education, diet counseling, and exercise guidance provided throughout the 12-week study period.

SUMMARY:
This clinical trial was conducted at the National Diabetes Center for Treatment and Research, Mustansiriyah University, Baghdad (Sept 2024-May 2025).

It evaluated the effect of mangosteen supplementation (500 mg twice daily) as an adjunct to sitagliptin/metformin (50/1000 mg twice daily) in newly diagnosed Type 2 Diabetes Mellitus (T2DM) patients over a period of 12 weeks.

* Sample: 47 patients completed the study (22 in sitagliptin/metformin group; 25 in sitagliptin/metformin + mangosteen group).
* Design: Prospective, randomized, controlled, open-label trial.
* Intervention: Both groups also received lifestyle modification (diet, exercise, diabetes education).
* Endpoints: Anthropometric measures, glycemic control (FBG, HbA1c, insulin, HOMA-IR, HOMA-B), lipid profile, oxidative stress (SOD1), inflammatory marker (IL-6), liver & kidney function, and safety monitoring.
* Statistical Analysis: Parametric/non-parametric tests, correlations, regression, and ANCOVA to assess changes and adjust for confounders.

DETAILED DESCRIPTION:
1. Patients

   * Inclusion: Adults (>30 years) with T2DM (AACE criteria), HbA1c 7.5-9%.
   * Exclusion: T1DM, insulin users, patients with complications, liver/kidney disease, other metabolic/endocrine disorders, patients on steroids/contraceptives/thyroid meds/supplements, pregnant/lactating women.
   * Ethics: Approved by Mustansiriyah University Ethics Committee. Written informed consent obtained.
2. Study Design

   * Type: Interventional, prospective, randomized, controlled, open-label.
   * Groups:
   * Group 1 (n=22): Sitagliptin/metformin 50/1000 mg twice daily + lifestyle modification.
   * Group 2 (n=25): Sitagliptin/metformin 50/1000 mg twice daily + Mangosteen 500 mg twice daily + lifestyle modification.
   * Duration: 12 weeks.
   * Compliance: Monitored via pill counts, phone follow-ups, monthly clinic visits.
3. Interventions & Protocol

   * All patients received standardized diabetes education and counseling.
   * Two-week washout for lipid-lowering drugs before enrollment to avoid confounding.
   * Data collected: demographics, socioeconomic, comorbidities, medication use, family history.
4. Measurements

   * Anthropometry: Weight, height, BMI, waist circumference, index of central obesity (ICO).
   * Samples:
   * Blood: Collected after 12-hour fasting (baseline & after 12 weeks). Serum separated for immediate and stored analysis.
   * Urine: Albumin/creatinine ratio to exclude nephropathy.
   * Biochemical tests:
   * Glycemic control: HbA1c (immunoassay), fasting blood glucose (hexokinase method), fasting serum insulin (ECLIA).
   * Insulin resistance & β-cell function: HOMA-IR, HOMA-B formulas.
   * Lipid profile: TC, HDL-C, TG, LDL-C, VLDL-C.
   * Inflammatory marker: Interleukin-6 (ELISA).
   * Oxidative stress marker: Superoxide dismutase-1 (ELISA).
   * Kidney function: Serum urea, creatinine, urinary ACR.
   * Liver function: AST, ALT, ALP.
5. Statistical Analysis

   * Software: SPSS v25.
   * Tests Used:
   * Normality: Shapiro-Wilk test.
   * Between-group: Independent t-test or Mann-Whitney U.
   * Within-group: Paired t-test or Wilcoxon signed-rank.
   * Categorical: Chi-square or Fisher's exact.
   * Correlations: Pearson test.
   * Regression: Linear regression for predictors of HbA1c change.
   * ANCOVA: Adjusted analysis for differences between groups (e.g., baseline HOMA-IR).
   * Significance: p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥30 years.
* Diagnosed with Type 2 Diabetes Mellitus according to American Association of Clinical Endocrinologists (AACE) criteria.
* HbA1c between 7.5% and 9%.

Exclusion Criteria:

* T1DM patients were excluded from study.
* T2DM patients receiving any anti-diabetic treatment other than the study intervention or T2DM patients receiving insulin therapy.
* Patients with T2DM complications or having liver disease, kidney disease.
* Patients with other metabolic diseases (thyroid disorders, adrenal disorders, growth hormone disorders and pituitary disorders) that may affect glycemic and metabolic status.
* Patients receiving drugs (steroids, contraceptives, anticoagulants and thyroid medications) or using other nutritional supplements or herbal remedies that may interfere with lab results.
* Pregnant or lactating women.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) | baseline and after 12 weeks
  HbA1c level will be measured using an immunoassay method (Roche Cobas c111 system) to assess glycemic control.

SECONDARY OUTCOMES:
Change in HOMA-IR (Insulin Resistance Index) | baseline and 12 weeks
  Calculated using fasting glucose and fasting insulin levels
Change in Fasting Blood Glucose (FBG) | Baseline and 12 weeks
  Measured by enzymatic hexokinase method (Roche Cobas c111 analyzer)
Change in HOMA-B (β-cell Function Index) | Baseline and 12 weeks
  Calculated using fasting insulin and fasting glucose concentrations
Change in Lipid Profile (TC, LDL-C, HDL-C, TG, VLDL-C) | Baseline and 12 weeks
  Measured by enzymatic colorimetric methods (Roche Cobas c111)
Change in Serum Interleukin-6 (IL-6) | Baseline and 12 weeks
  Measured by ELISA (sandwich principle)
Change in Serum Superoxide Dismutase-1 (SOD1 | Baseline and 12 weeks
  Measured by competitive ELISA kit
Change in Liver Enzymes (AST, ALT, ALP) | Baseline and 12 weeks
  Measured by Roche Cobas c111 analyzer
Change in Kidney Function (Serum Creatinine, Urea, and Urinary ACR) | Baseline and 12 weeks
  Measured by Roche Cobas c111 analyzer and Combilyzer 13 system

CONTACTS AND LOCATIONS:
Overall Officials: Manal Kh Abdulridha, Prof., Principal Investigator — Department of Clinical Pharmacy, College of Pharmacy, Mustansiriyah University
Locations (1):
- National Diabetes Center for Treatment and Research, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Only aggregated results and statistical analyses will be published in scientific journals or presented at conferences.